CLINICAL TRIAL: NCT06882408
Title: Evaluation of the Photorefraction Screener Snapsight in Comparison With Cycloplegia Table-top Autorefractor in Ametropia in Pediatric Population Between 3 and 8yo, Multicenter French Study.
Brief Title: The Objective of This Study is to Evaluate the Perfomance of a Photorefraction Device for Screening Ametropia in Children. Eligible Participants Will Undergo Multiple Refractive Error Measurements, Visual Acuity and Strabismus Assessments During a Single Evaluation Visit.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WS10386-EPSS; 2024-A00780-47 (Other: ANSM)
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Ametropia; Myopia; Refractive Error; Myopia; Astigmatism
MeSH Terms: conditions — Refractive Errors; Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Snapsight photorefraction device (Experimental)
  Interventions: Device: Photorefraction device under investigation; Device: Comparator device, Tabletop auto-refractometer; Device: Comparator device, portable photorefraction device; Other: Distance visual acuity assessments; Other: Subjective refraction and far visual acuity; Other: Strabismus assessment

INTERVENTIONS:
Device: Photorefraction device under investigation — Objective refraction measurement with and without cyclopegia
Device: Comparator device, Tabletop auto-refractometer — Objective refraction measurement with and without cyclopegia
Device: Comparator device, portable photorefraction device — Objective refraction measurement with and without cyclopegia
Other: Distance visual acuity assessments — Distance visual acuity is assessed with the refraction measures found by the device under investigation and the comparator device with and without cyclopegia.
Other: Subjective refraction and far visual acuity — Subjective refraction is assessed and far visual acuity is assessed with the found refraction measures
Other: Strabismus assessment — Strabismus is assessed with the refraction measures found by the device under investigation and the comparator device with and without cyclopegia.

SUMMARY:
The goal of this clinical trial is to evaluate the performance of a photorefraction screener in terms of sensibility, sensitivity and accuracy on children aged 3 to 8 y.o. The main objectives of the study are:

* Evaluate the performances of the device in comparison with the gold standard, i.e. a tabletop refractometer.
* Assess the agreement of the measures obtained with the device with those obtained with the gold standard.

DETAILED DESCRIPTION:
Participants after verification of their eligibility and informed consent, participate to a single evaluation visit during which several objective refraction measurements are performed with the investigational device, a tabletop refractometer and a comparable vision screener with and without cyclopegia. Additionally far vision visual acuity, strabismus assessments and subjective refraction measurement are also performed by investigators.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 3-8 years when included in the study
* All skin phototypes (I to VI according to the Fitzpatrick classification)
* Wearing glasses or not
* Capacity to give valid consent
* Capacity to follow the protocol to obtain reliable measure
* Under French medical insurance

Exclusion Criteria:

* Under myopia control solution that may have an impact on refractive error (such as: atropine, orthokeratology,..)
* Wearing contact lenses
* Ocular or systemic pathology that may have an impact on vision or may interfere with the study measures (except strabismus)
* Under medication that may have an impact on vision or may interfere with study measurements
* Known contraindication to the active substance or to one of the excipients of eye drops (Mydriaticum 0.5%, Skiacol 0.5%)
* Known risk of angle-closure glaucoma
* Participation to another study that may have an impact on vision or may interfere with the study measures

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 315 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Perfomance evaluation for ametropia screening | One day (all measurements are taken during a single evaluation visit).
  The performance of the device in terms of sensitivity is evaluated by comparison with a tabletop refractometer.

SECONDARY OUTCOMES:
Agreement of refraction measurements obtained with the device under investigation and a tabletop refractometer | One day (all measurements are taken during a single evaluation visit).
  The evaluated refraction measurements are the spherical equivalent and Jackson's cylindrical vectors.
Perfomance evaluation for ametropia screening | One day (all measurements are taken during a single evaluation visit).
  The performance of the device in terms of sensitivity, specificity, positive and negative predictive values are evaluated by comparison with a tabletop refractometer.
Perfomance evaluation for amblyopia screening | One day (all measurements are taken during a single evaluation visit).
  The performance of the device in terms of sensitivity, specificity, positive and negative predictive values are evaluated by comparison with a tabletop refractometer or the masking test and prism bars for strabismus.
Safety assessment and device failures | One day (all measurements are taken during a single evaluation visit).
  Type, frequency and severity of adverse events and device failures are evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Aranaud Sauer, MD, PhD, FEBO, Principal Investigator — Hôpital Civil de Strasbourg
Locations (2):
- France (2):
  - Dr Krafft private practice, Nancy, France
  - Hôpital civil de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No